CLINICAL TRIAL: NCT07185906
Title: The Effect of WhatsApp-Based Education and Counseling on Breastfeeding Self-Efficacy, Body Satisfaction, Healthy Lifestyle Behaviors, and Weight Retention in Postpartum Women: A Randomized Controlled Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Inonu University (Other)
Responsible Party: Principal Investigator, FİGEN BİLGİN, PhD Candidate in Women's Health and Diseases Nursing, Inonu University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: IU-SBE-FB-01
Record Dates: First submitted 2025-09-15; First posted 2025-09-22 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2024-06

CONDITIONS: Post Partum; Breast Feeding; Body Image; Health Behavior; Weight Change; Postpartum Period
MeSH Terms: conditions — Breast Feeding; Health Behavior; Body Weight Changes | interventions — Educational Status

STUDY DESIGN:
Intervention Model Description: Participants were randomly assigned to intervention and control groups in a parallel design.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental: WhatsApp-based Education and Counseling (Experimental): Participants receive an 8-week WhatsApp-based education and counseling program in addition to routine postpartum care. The intervention includes short educational videos, weekly messages, and feedback provided through WhatsApp. Content covers breastfeeding techniques, recognition of infant hunger cues, milk expression and storage, management of common breastfeeding problems, healthy nutrition, body satisfaction, and postpartum weight management.
  Interventions: Behavioral: education
- Control Group (No Intervention): Participants receive routine postpartum care provided by Family Health Centers. They do not receive any structured WhatsApp-based education or counseling.

INTERVENTIONS:
Behavioral: education — WhatsApp-based training was provided
  Arms: Experimental: WhatsApp-based Education and Counseling

SUMMARY:
Brief Summary:

This randomized controlled trial aimed to evaluate the effect of WhatsApp-based education and counseling on breastfeeding self-efficacy, body satisfaction, healthy lifestyle behaviors, and weight retention in postpartum women. The study was conducted between January and March 2025 at four Family Health Centers in Siirt, Turkey. A total of 120 postpartum women were randomly assigned to the intervention and control groups. The intervention group received an 11-week WhatsApp-based education program, including short videos and counseling sessions prepared under the guidance of the Health Promotion Model. Data were collected at baseline, 3 months, and 6 months using validated instruments: the Postnatal Breastfeeding Self-Efficacy Scale, the Body Satisfaction Scale, and the Health-Promoting Lifestyle Profile II. The primary outcomes were breastfeeding self-efficacy and body satisfaction, while secondary outcomes included healthy lifestyle behaviors and postpartum weight retention. The findings are expected to provide evidence for the effectiveness of mobile health interventions in improving maternal health outcomes during the postpartum period.

ELIGIBILITY:
Inclusion Criteria:

* • Women in the postpartum period (within the first week after delivery)

  * Aged 18-49 years
  * Able to read and understand Turkish
  * Owning a smartphone with internet access and WhatsApp installed
  * Willing to participate in the study and provide informed consent

Exclusion Criteria:

* Women with medical complications that prevent breastfeeding (e.g., serious maternal illness, contraindications to breastfeeding)

  * Infants with conditions that prevent breastfeeding (e.g., congenital anomalies affecting sucking or swallowing)
  * Women with severe psychiatric disorders or cognitive impairments that may interfere with participation
  * Women who do not agree to participate or withdraw consent during the study

Ages: 18 Years to 49 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Only postpartum women are eligible to participate in this study.
Enrollment: 86 (Actual)
Dates: Start 2025-01-01 (Actual); Primary Completion 2025-06-30 (Actual); Study Completion 2025-07-30 (Actual)

PRIMARY OUTCOMES:
Breastfeeding Self-Efficacy, | Baseline, 3 months postpartum, 6 months postpartum
  The Postnatal Breastfeeding Self-Efficacy Scale will be used to assess mothers' confidence and self-efficacy in breastfeeding practices. Changes in mean scores between groups and over time will be evaluated.
Body Satisfaction | Baseline, 3 months postpartum, 6 months postpartum
  The Body Satisfaction Scale will be used to measure mothers' satisfaction with their body image during the postpartum period. Changes in scores across intervention and control groups will be compared.

SECONDARY OUTCOMES:
Healthy Lifestyle Behaviors | Baseline, 3 months postpartum, 6 months postpartum
  Health-promoting lifestyle behaviors will be measured using the Health-Promoting Lifestyle Profile II (HPLP-II). Total and subscale scores (nutrition, physical activity, stress management, interpersonal relations, health responsibility, and spiritual growth) will be analyzed.
Postpartum Weight Retention | Baseline, 3 months postpartum, 6 months postpartum
  Postpartum weight retention will be calculated by subtracting the pre-pregnancy weight from the mother's postpartum weight at each measurement time. Changes will be compared between intervention and control groups.

CONTACTS AND LOCATIONS:
Locations (1):
- ): Inonu University, Faculty of Health Sciences, Siirt, Siirt, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
The individual participant data will not be shared. Only aggregated results will be published in scientific journals.

REFERENCES:
- See also: Related Info — https://www.inonu.edu.tr